CLINICAL TRIAL: NCT06755138
Title: Research on the Relationship Between Scoliosis, Pain, Quality of Life, and Trunk Muscle Compensation Patterns During Functional Upper Extremity Movements Among Patients with Duchenne Muscular Dystrophy Using Surface Electromyography and Computer Vision Analysis.
Brief Title: Research on the Relationship Between Scoliosis, Pain, Quality of Life, and Trunk Muscle Compensation Patterns Among Patients with Duchenne Muscular Dystrophy.
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Woo Hyung Lee, Associate professor, Seoul National University Hospital
Other Study IDs: 0420240390
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- DMD group: Duchenne muscular dystrophy group for analysis
  Interventions: Other: Observational Assessment
- Healthy control group: Healthy age-matched group to compare scoliosis, upper limb function level, pain, quality of life, and trunk muscle compensation patterns using sEMG and computer vision
  Interventions: Other: Observational Assessment

INTERVENTIONS:
Other: Observational Assessment — This study includes the use of surface electromyography (sEMG), video analysis, and questionnaires to assess trunk compensation patterns and their relationship with scoliosis, functional, quality-of-life, and pain parameters

SUMMARY:
* Objective:

The objective of this observational study is to evaluate and quantify trunk muscle compensatory movement patterns in patients with Duchenne Muscular Dystrophy (DMD) using computer vision technology. Additionally, the study seeks to explore the relationship between these compensatory patterns and scoliosis, upper limb function, pain levels, and quality of life during functional upper limb movements.

* Key Research Questions:

  1) Can trunk compensatory movement patterns be accurately measured using computer vision analysis? 2) Are these compensatory patterns correlated with scoliosis, upper limb function levels, pain, and quality of life? 3) Do these patterns and their correlations change over time?
* Methodology:

  1. Participants: Patients diagnosed with Duchenne Muscular Dystrophy will be recruited for this study.
  2. Assessments:
* Scoliosis Evaluation:

  1. Cobb angle measurement via X-ray imaging.
  2. Upper Limb Function Assessment:
  3. Performance of the Upper Limb Module 2.0 (PUL 2.0).
  4. Brooke Upper Extremity Functional Classification Score.
  5. Korean version of the Duchenne Muscular Dystrophy Functional Ability Self-Assessment Tool (K-DMDSAT).
* Pain Measurement:

  1. Korean version of the PainDETECT Questionnaire (KPD-Q).
  2. Short Form McGill Pain Questionnaire.
  3. Quality of Life Assessment:
* Duchenne Muscular Dystrophy Quality of Life Questionnaire (DMD-QoL).

  1. Trunk Compensation Analysis:
* Surface electromyography (sEMG) to measure muscle activation.
* Video analysis using computer vision to quantify trunk compensatory movement patterns.
* The following tasks will be evaluated using the dominant arm for sEMG and video analysis:

  i. Pouring water into a cup. ii. Lifting a cup to drink water. iii. Grooming the front of the hair. iv. Moving small blocks within one minute (Box and Block Test). v. Reaching toward nearby objects in the front, left, and right directions.
* Front: Directly in front of the participant's line of sight.
* Left and right: Approximately 45 degrees to the left and right from the participant's front.
* Nearby objects: A water bottle or cup weighing approximately 250g, placed at arm's length.

vi. Reaching toward distant objects in the front, left, and right directions.

* Distant objects: A water bottle or cup weighing approximately 250g, placed at 1.5 times the participant's arm length.
* The sEMG attachment sites are as follows:

  i. Muscles for assessing upper limb functional movements:
  1. Deltoid
  2. Pectoralis major
  3. Trapezius
  4. Biceps brachii ii. Muscles for assessing trunk compensatory actions:

  <!-- -->

  1. Sternocleidomastoid
  2. Longissimus muscle
  3. External oblique abdominal muscle

ELIGIBILITY:
1. Inclusion Criteria (1) Duchenne Muscular Dystrophy (DMD) Group

   * Individuals with a confirmed genetic diagnosis of Duchenne Muscular Dystrophy.
   * Aged over 10 years but under 30 years.
   * Brooke Scale score between 2 and 5.
   * Shoulder abductor muscle strength below grade 3 on the Manual Muscle Test (MMT).

     (2) Healthy Control Group
   * Individuals with no history or current diagnosis of musculoskeletal or neuromuscular disorders.
   * Aged over 10 years but under 30 years.
   * Shoulder muscle strength of grade 4+ or higher on the Manual Muscle Test (MMT).
   * Individuals capable of understanding a detailed explanation of the study procedures and voluntarily providing written informed consent.
2. Exclusion Criteria (1) Duchenne Muscular Dystrophy (DMD) Group

   * Individuals unable or unwilling to provide informed consent.
   * Brooke Scale score of 1 or 6.
   * Severe cognitive impairment preventing the performance of simple tasks. (2) Healthy Control Group
   * Individuals unable or unwilling to provide informed consent.
   * Shoulder muscle strength of grade 4 or lower on the Manual Muscle Test (MMT).

Ages: 11 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study will recruit participants from two populations: individuals with Duchenne Muscular Dystrophy (DMD) and age-matched healthy controls. The DMD group includes subjects aged 10-30 years with a confirmed genetic diagnosis, Brooke Scale scores of 2-5, and shoulder abduction strength below grade 3 on the Manual Muscle Test (MMT). These participants represent a population with progressive neuromuscular decline and compensatory trunk muscle activity. The healthy control group consists of subjects aged 10-30 years matched to recruited DMD groups, with no history of musculoskeletal or neuromuscular disorders and shoulder strength of grade 4+ or higher on the MMT. Both groups must understand study procedures and provide informed consent. This population ensures a meaningful comparison of trunk compensatory movement patterns between DMD patients and healthy individuals, offering valuable insights into functional adaptations and their implications for care.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Surface Electromyography (sEMG) | enrollment, 6 months after, and 12 months after since the enrollment
  The purpose of using surface electromyography (sEMG) in this study is to measure and analyze the activation levels and patterns of trunk compensatory muscles during the performance of functional upper limb movements. This assessment aims to understand how trunk muscles compensate for upper limb movements, particularly in relation to task performance efficiency.
Computer Vision-Based Video Analysis | enrollment, 6 months after, and 12 months after since the enrollment
  Videos are recorded simultaneously with surface electromyography (sEMG) while participants perform functional upper limb movements. Recordings are taken from two perspectives: the front view and the dominant arm side view, with synchronized matching of the videos. Video recording is conducted using a video camera mounted on a fixed tripod.
  The recorded videos are analyzed using a convolutional neural network (CNN)-based body part detection model, producing skeleton-based outputs for movement analysis. The relative trunk motion of the participant is extracted as positional coordinates over time, which are further processed to calculate velocity, acceleration, and jerk. These time-series signals are analyzed for smoothness and sample entropy. By matching the movement data with corresponding sEMG signals, biomechanical compensatory parameters are identified and key compensatory features are derived. Comparative analyses with healthy controls are performed to validate these parameters.

SECONDARY OUTCOMES:
Brooke Score | enrollment, 6 months after, and 12 months after since the enrollment
  The Brooke Score is a functional assessment tool specifically designed to evaluate upper limb abilities in patients with Duchenne Muscular Dystrophy (DMD). An occupational therapist or physical therapist instructs participants to perform specific movements, and the assessment is based on the participant's ability to successfully complete these tasks.
  The scale ranges from 1 to 6, with lower scores indicating better upper limb function
Performance of the Upper Limb Module 2.0 (PUL 2.0) | enrollment, 6 months after, and 12 months after since the enrollment
  A functional scale specifically designed to evaluate upper limb abilities in patients with Duchenne Muscular Dystrophy (DMD), assessed by an occupational or physical therapist. It consists of 22 items divided into three levels: shoulder level (6 items, maximum score 12), mid-level (9 items, maximum score 17), and distal level (7 items, maximum score 13), with a total possible score of 44. Each level is scored separately, and participants are instructed to perform specific tasks, with their performance evaluated accordingly.
Korean version of the Duchenne Muscular Dystrophy Functional Ability Self-Assessment Tool (K-DMDSAT) | enrollment, 6 months after, and 12 months after since the enrollment
  A patient-reported outcome measure designed to evaluate and describe the functional status of individuals with Duchenne Muscular Dystrophy (DMD) across the disease progression. It comprises four domains: arm function, walking, mobility, and respiratory support. Patients are asked to select the most difficult task they can still perform. The tool demonstrates excellent reliability, with inter-rater and test-retest reliability scores (ICC 0.958 and 0.987, respectively). Scoring ranges from 0-8 for arm function and walking, 0-10 for mobility, and 0-2 for respiratory support, with a total maximum score of 28.
Korean version of the PainDETECT Questionnaire (KPD-Q) | enrollment, 6 months after, and 12 months after since the enrollment
  A tool developed to assess neuropathic pain and is also applicable for evaluating other types of pain. It evaluates four domains: pain intensity, location, pattern, and radiating pain, with a total maximum score of 38. Based on the score, pain can be classified into nociceptive pain, unclear pain, or neuropathic pain categories
Short Form McGill Pain Questionnaire (SF-MPQ) Korean version | enrollment, 6 months after, and 12 months after since the enrollment
  a self-reported tool designed to assess both the quality and intensity of subjective pain. It includes 11 adjectives describing the sensory aspects of pain and 4 adjectives related to its emotional impact. Participants also rate their current pain intensity on a scale from 0 (no pain) to 5 (worst possible pain) and indicate the overall intensity of their pain on a 10 cm visual analog scale (VAS).
Duchenne Muscular Dystrophy Quality of Life Questionnaire (DMD-QoL) | enrollment, 6 months after, and 12 months after since the enrollment
  Specifically designed to reflect the unique needs and experiences of individuals with Duchenne Muscular Dystrophy (DMD). It comprises 14 items across key domains, including physical health, emotional well-being, social functioning, school and academics, pain and symptom management, and independence and autonomy. Participants respond using a Likert scale to indicate the degree of agreement or frequency for each item. While the questionnaire is intended to be self-reported, caregivers or guardians may complete it on behalf of the patient if age or cognitive function limits independent completion.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No